CLINICAL TRIAL: NCT02600078
Title: The Evaluation of a Mobile Device to Measure Ataxia With High Altitude Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Sports Medicine Research Foundation (Other)
Responsible Party: Principal Investigator, Elliott Boake, Masters of Science Student, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H15-02093
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Hypoxia
Keywords: hypoxia; ataxia
MeSH Terms: conditions — Hypoxia; Ataxia | interventions — Heart Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate Hypoxia (Active Comparator): Subjects will be exposed to moderate hypoxia and measures of balance, heart rate, pulse oxygen saturation, questionnaires, and coordination tasks will be examined at set time intervals during the hypoxic exposure.
  Interventions: Device: AMS Monitor App; Other: Lake Louise Score; Other: Balance Error Scoring System; Other: Heart Rate & Pulse Oxygen Saturation
- Sham (Sham Comparator): Subjects will be exposed to sham and measures of balance, heart rate, pulse oxygen saturation, questionnaires, and coordination tasks will be examined at set time intervals during the hypoxic exposure.
  Interventions: Device: AMS Monitor App; Other: Lake Louise Score; Other: Balance Error Scoring System; Other: Heart Rate & Pulse Oxygen Saturation
- Mild Hypoxia (Active Comparator): Subjects will be exposed to mild hypoxia and measures of balance, heart rate, pulse oxygen saturation, questionnaires, and coordination tasks will be examined at set time intervals during the hypoxic exposure.
  Interventions: Device: AMS Monitor App; Other: Lake Louise Score; Other: Balance Error Scoring System; Other: Heart Rate & Pulse Oxygen Saturation

INTERVENTIONS:
Device: AMS Monitor App — Participants will complete a novel coordination task performed on an android phone.
Other: Lake Louise Score — Participants will complete a questionnaire to assess acclimatization to hypoxia.
Other: Balance Error Scoring System — Participants will complete a series of static stance positions to evaluate their ability to maintain balance.
Other: Heart Rate & Pulse Oxygen Saturation — Participants will have their heart rate and pulse oxygen saturation continuously monitored throughout the entire exposure.

SUMMARY:
With exposure to high altitude some individuals will develop acute mountain sickness (AMS). Current evaluation of AMS can make it difficult to rule out other possible conditions. Evaluation of ataxia, as measured by the performance of a coordinated task, can aide in the correct diagnosis of AMS. The investigators have developed novel finger-tapping tasks on a mobile device to assess both reaction time and accuracy. The proposed research will evaluate the utility of this tool in assessing human acclimatization to hypoxia.

DETAILED DESCRIPTION:
Introduction: Hypoxia is the reduction in partial pressure of oxygen that occurs with exposure to altitude. Individuals acclimatize at different rates and to different degrees meaning that those who are slow to make the necessary physiological adjustments will develop signs and symptoms of acute mountain sickness (AMS). AMS is marked by headache, gastrointestinal disturbances, insomnia, fatigue and ataxia, which can be evaluated using subjective questionnaires such as the Lake Louise Score (LLS). Evaluation of AMS by solely using subjective questionnaires can make differential diagnosis of other possible pathologies difficult. Ataxia is characterized by poor coordination in the absence of significant weakness. Ataxia can be assessed with the performance of a coordinated task. The investigators have developed a novel finger-tapping task on a mobile device to assess both reaction time and accuracy. The proposed research will evaluate the utility of this tool in assessing human acclimatization to hypoxia, which could ultimately serve as a novel, objective methodology in the diagnosis of AMS.

Hypothesis: (1) When exposed to simulated altitude (equivalent to 4200m above sea level), subjects will exhibit diminished coordination relative to a sham exposure. (2) Reaction time of novel coordination tasks will positively correlate with heart rate, balance, and LLS. (3) Accuracy of novel coordination tasks will negatively correlate with heart rate, balance, and LLS.

Methods: A repeated-measures design with a familiarization trial, a hypoxic trial, and a sham trial will be used. Sixteen healthy adults will be exposed to normobaric hypoxia in the investigator's chamber, simulating an elevation of 4200m above sea level. Subjects will be measured for pulse oxygen saturation, heart rate, and will complete the LLS, the Balance Error Scoring System (BESS), as well as two electronic finger tap coordination tasks prior to, and at 5 minutes, 4, and 12 hours into the altitude chamber exposure.

Outcomes: This research will enhance the investigators understanding of the relationship between coordination, balance, and acclimatization to hypoxia. It will allow us to validate a new objective tool in the measurement of acclimatization with exposure to hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female Gender
* Minimum Age of 18 years
* Maximum Age of 45 years
* Have not traveled to an altitude of 3000m or higher in 3 months prior to testing
* No history of migraines or concussion
* Not Smokers
* Females must be using monophasic birth control
* Not easily claustrophobic
* English Speaking

Exclusion Criteria:

* Non-English speaking individuals
* Subjects younger than 18 years old or older than 45 years old
* Subjects who visit an altitude of 3000m or greater within three months prior to the study
* Subjects with a history of cardiovascular or pulmonary conditions such as; uncontrolled congestive heart failure, COPD, pulmonary hypertension, or sickle cell disease
* Subjects with a history of migraines or concussion
* Smokers
* Females not using monophasic birth control pills
* Subjects experiencing withdrawal symptoms due to abstinence from caffeine
* Easily claustrophobic individuals

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in score of a coordination test. | Coordination test will be taken at baseline and at 5 minutes, 4 and 12 hours into a simulated altitude exposure.

SECONDARY OUTCOMES:
Change in severity of symptoms based on questionnaire. | Symptoms questionnaire will be assessed at baseline and at 5 minutes, 4 and 12 hours into a simulated altitude exposure.
Change in score of a balance test. | Balance test will be taken at baseline and at 5 minutes, 4 and 12 hours into a simulated altitude exposure.
Change in heart rate. | Heart rate will be assessed at baseline and at 5 minutes, 4 and 12 hours into a simulated altitude exposure.
Change in pulse oxygen saturation | Pulse oxygen saturation will be assessed at baseline and at 5 minutes, 4 and 12 hours into a simulated altitude exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Koehle, MD, Principal Investigator — University of British Columbia
Locations (1):
- Environmental Physiology Laboratory, Vancouver, British Columbia, Canada